CLINICAL TRIAL: NCT06973083
Title: Efficacy and Safety of Robot-assisted Endoscopic Submucosal Dissection for Colorectal Neoplasm: A Randomized Controlled Trial.
Brief Title: Efficacy and Safety of Robot-assisted Endoscopic Submucosal Dissection for Colorectal Neoplasm
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Xiuli Zuo, Professor, MD, PhD, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: QLCR20230523
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Robot Surgery; Endoscopic Submucosal Dissection (ESD); Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FASTER-assisted ESD (Experimental): Patients in this group undergo ESD with the assistance of the FASTER system.
  Interventions: Procedure: FASTER-assisted ESD
- Conventional ESD (Active Comparator): Patients in this group undergo ESD following the clinically established pattern.
  Interventions: Procedure: Conventional ESD

INTERVENTIONS:
Procedure: FASTER-assisted ESD — The patients who are randomly assigned to the FASTER-assisted ESD group will undergo the ESD procedure with the assistance of the FASTER system.
  Arms: FASTER-assisted ESD
Procedure: Conventional ESD — The patients who are randomly assigned to the conventional ESD group will undergo the ESD following the clinically established pattern.
  Arms: Conventional ESD

SUMMARY:
The objective of this study is to investigate the role of the flexible auxiliary single-arm transluminal endoscopic robot (FASTER) system in colorectal endoscopic submucosal dissection (ESD) and to validate its superiority over conventional ESD in terms of reducing procedural difficulty, shortening procedure time, and enhancing procedural safety.

The main questions it aims to answer are:

Does the use of the FASTER system improve the dissection speed of the ESD procedure? Does the use of the FASTER system reduce the procedure and dissection time, improving the efficacy of the ESD procedure? Does the use of the FASTER system reduce the rate of perforation and hemorrhage, improving the safety of the ESD procedure? Researchers will compare FASTER-assisted ESD and conventional ESD to evaluate the safety and efficacy of the FASTER system.

Participants will:

Be randomly assigned to the group with ESD using the traditional procedure or to the group with ESD assisted by the FASTER system.

Keep a diary of their symptoms after the procedure. ESD has gained widespread acceptance as the standard method for treating early-stage gastrointestinal cancers. However, ESD is a technically demanding and intricate procedure that requires advanced proficiency of operators, with a heightened risk of complications such as hemorrhage and perforation. The inherent challenges of the colorectal ESD are further amplified by the thin mucosa, highly tortuous and flexible lumen, and occasional obstruction of lesions by mucosal folds, all of which collectively elevate both the procedural difficulty and the probability of postoperative complications. Adequate exposure of the submucosa layer through effective tissue traction is vital for the safe and effective performance of ESD. The FASTER system is designed to overcome this technical difficulty.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-85.
* Patients with pathologically verified colorectal neoplasms scheduled to undergo ESD.

Exclusion Criteria:

* Patients have lesions with confirmed or potential deep submucosal invasion or lymph node metastasis or other conditions that are not suitable for endoscopic therapy.
* Patients with severe underlying diseases precluding endotracheal intubation, general anesthesia, or surgery.
* Patients have a history of colorectal malignancy with previous radiotherapy or operative treatment leading to changes in colorectal structure.
* Patients have lesions with local recurrence after endoscopic resection.
* Patients unable to obtain informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
procedure time | Within 24 hours after the procedure.
  Procedure time is the time from the beginning of injection to the completion of dissection.

SECONDARY OUTCOMES:
dissection time | Within 24 hours after the procedure.
  Dissection time is the time from the beginning of dissection to the completion of dissection.
dissection speed | Within 24 hours after the procedure.
  Dissection speed is defined as the lesion area divided by the dissection time.
en bloc resection rate | Within 24 hours after the procedure.
  En bloc dissection refers to the complete removal of the entire lesion in a single piece.
R0 resection rate | Within 24 hours after the procedure.
  R0 resection is defined as en bloc resection with negative vertical and horizontal margins.
perforation rate | Within 24 hours after the procedure.
  Perforation were defined as: endoscopic visualization of mural transection during ESD, or postoperative clinical signs combined with radiologically confirmed pneumoperitoneum.
postoperative hemorrhage rate | Within 24 hours after the procedure.
  Post-ESD hemorrhage was strictly defined as meeting ≥1 of: hematemesis or melena with dizziness, hemoglobin decline >20 g/L, SBP drop >20 mmHg or HR elevation >20 bpm, presence of bloody fluid in nasogastric tube drainage, or active bleeding confirmed by repeat endoscopy.
intraoperative hemorrhage rate | Within 24 hours after the procedure.
the proportion of intraoperative hemorrhage ≥ grade 2 | Within 24 hours after the procedure.
  Intraoperative hemorrhage is divided into four grades: Grade 0 means no significant bleeding is observed during the procedure. Grade 1 means minimal bleeding, which could stop spontaneously or be easily controlled by cauterization with a dual knife. Grade 2 refers to minor hemorrhage that requires multiple cauterizations with a dual knife or hemostatic forceps. Grade 3 indicates massive hemorrhage that requires multiple cauterizations with hemostatic forceps.
hemostasis time | Within 24 hours after the procedure.
  Hemostasis time referred to the time from the detection of submucosal bleeding until hemostasis was completed.
muscular injury rate | Within 24 hours after the procedure.
  Muscular injury is described as visible damage to the muscularis propria.
direct-vision dissection rate | Within 24 hours after the procedure.
  Direct-vision dissection time is the time that the endoscopist can directly observe the tip of the dual knife and the submucosal layer at the same time. By dividing the direct-vision dissection time by the total dissection duration, the direct-vision dissection rate is calculated.
postoperative pain score | 3 days after the procedure.
  Postoperative pain score was assessed via the 11-point Numerical Rating Scale (NRS: 0=no pain, 10=worst imaginable pain). Patients independently rated their pain intensity on postoperative day 3, with scores categorized as mild (1-3), moderate (4-6), or severe (7-10).*
the frequency of supplemental injections | Within 24 hours after the procedure.
  Supplemental injection refers to injections performed after the beginning of the dissection.
the supplemental injections time | Within 24 hours after the procedure.
  The time of supplementary injection is from the insertion of the injection needle into the submucosal layer until the injection is completed and the needle is withdrawn.
Volume of injection fluid used in supplemental injections | Within 24 hours after the procedure.
the frequency of intraoperative patient positioning changes | Within 24 hours after the procedure.
time required for patient positioning changes | Within 24 hours after the procedure.
NASA-TLX scale scores | Within 24 hours after the procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China